CLINICAL TRIAL: NCT04337840
Title: Analysis on the Infection Risk, Prognosis, and Drug Sensitivity of Klebsiella Pneumoniae.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202003047RINA
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-03

CONDITIONS: Klebsiella Pneumoniae Sepsis
Keywords: risk factors ,outcomes,Drug Susceptibility,Klebsiella pneumoniae

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Nosocomial infections are increasing rapidly both internationally and domestically, especially carbapenem-resistant Klebsiella pneumoniae infections. However, there were still lack of evidence about the risk and prognosis in Taiwan. The choice of drug and related sensitivity test was also limited. We would analyze the infection risk, prognosis, and drug sensitivity of Klebsiella pneumoniae and focus on strategy to manage carbapenem-resistant Klebsiella pneumoniae infections.

ELIGIBILITY:
All adult patients (≥18 years) with K. pneumoniae bloodstream infection were included. Patients were excluded if there was other recognized bacteremia within two weeks before or after the first episode of K. pneumoniae bloodstream infection.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted at the National Taiwan University Hospital (NTUH), a medical center with 2400 beds in Taipei City. We studied patients with K. pneumoniae bloodstream infection between October 2017 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-05 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
All-cause 28-day mortality | 2017-2019

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chung Chuang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan